CLINICAL TRIAL: NCT01001520
Title: Neural Substrates of Cognitive Deficits in Nicotine Withdrawal
Brief Title: Neural Substrates in Nicotine Withdrawal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 809858; R01DA026849 (NIH)
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-05

CONDITIONS: Tobacco Use Disorder
Keywords: Genetics; Nicotine; Cognition; fMRI
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Sugar Pill) (Placebo Comparator): 11-day placebo-controlled medication period
  Interventions: Drug: Placebo
- Tolcapone (Active Comparator): 11-day phase, tapered dosing scheduled (Day 1: 100mg three times daily, Days 2-8: 200mg three times daily, Day 9: 200mg twice daily, Day 10: 200mg once daily, Day 11: 100mg once daily); oral dosing; medication is encapsulated by the University of Pennsylvania's Investigational Drug Service (IDS)
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Drug: Tolcapone — Participants will be asked to take study medication each day for both 11-day study medication periods.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take tolcapone during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by tolcapone during the second medication period.
  Other Names: Tasmar
  Arms: Tolcapone
Drug: Placebo — Participants will be asked to take study medication each day for both 11-day study medication periods.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take tolcapone during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by tolcapone during the second medication period.
  Arms: Placebo (Sugar Pill)

SUMMARY:
This study will test the hypothesis that a medication called tolcapone (Brand Name: Tasmar) will help reduce cognitive problems that smokers experience when they quit. This study will also determine whether the benefits of this medication differ depending on a smokers' genetic background.

DETAILED DESCRIPTION:
Tolcapone, an FDA-approved treatment for Parkinson's disease, improves cognitive performance in healthy controls with COMT val/val genotypes, putatively by increasing prefrontal dopamine levels. We propose a within-subject double-blind cross-over neuroimaging study of short-term (11 days) treatment with tolcapone (vs. placebo).

Thirty chronic smokers (15 with val/val genotypes and 15 with val/met or met/met genotypes) will undergo blood oxygenation level dependent (BOLD) fMRI during the two medication periods:

1. after 24 hours of monitored abstinence while on tolcapone, and
2. after 24 hours of monitored abstinence while on placebo (medication order counterbalanced with at least a 10-day washout).

The BOLD fMRI data will be acquired while subjects perform a working memory task (Fractal N-back), a sustained attention task (Continuous Performance Task; CPT), and a response inhibition task (Go/No-Go). The primary outcome is medication effects (within subject) on task-related BOLD activation after 24 hours of abstinence. Changes in behavioral performance and subjective symptoms will be examined in relation to brain activity changes.

The proposed study will provide a critical mechanistic understanding of the role of COMT in abstinence-induced cognitive symptoms that promote smoking relapse. Information obtained in this study may further establish cognitive performance measures as endophenotypes for nicotine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who are between 18 and 65 years of age who self-report smoking at least 10 cigarettes (menthol and non-menthol) per day for at least the last 6 months.
* Healthy as determined by the Study Physician, based on a medical evaluation including medical history and physical examination, psychiatric evaluation, and liver function tests (LFTs and GGT enzyme levels).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
* Women of childbearing potential must consent to use a medically accepted method of birth control while participating in the study (e.g., condoms and spermicide, oral contraceptive, Depo-provera injection, contraceptive patch, tubal ligation) and have 3 months of regular menstrual cycles.
* Capable of providing a Carbon Monoxide (CO) breath test reading greater than 10 parts per million (ppm) at the medical screening visit.

Exclusion Criteria:

Smoking behavior

* Current enrollment or plans to enroll in another research or smoking cessation program in the next 3 months.
* Provide a CO reading less than or equal to 10ppm at the medical screening visit.
* Plans to use nicotine substitutes (gum, patch, lozenge, e-cigarette) while enrolled in the study.

Alcohol/Drug Exclusion:

* History (past 2 years) or current diagnosis of substance abuse and/or currently receiving treatment for substance abuse (alcohol, THC, cocaine, PCP, amphetamines, methamphetamines, MDMA/ecstasy, opiates, methadone, benzodiazepines, tricyclic antidepressants, and barbiturates).
* Current alcohol consumption that exceeds 21 standard drinks/week over the last 6 months.
* Positive urine drug screen (for substances listed previously) at the medical screening visit or either testing day.
* Breath Alcohol Concentration (BrAC) assessment greater than or equal to 0.01 at medical screening visit or either testing day.

Medication Exclusion Criteria:

Current use or recent discontinuation (within last 28 days) of any medication including the following:

* Any form of psychotropic medications including: Antipsychotics; Mood-stabilizers (e.g., lithium, valproic acid, carbamazepine/tegretol); Anti-depressants (tricyclics, SSRI's, MAOI's, non-selective MAOIs, Wellbutrin, St. John's Wort); Anti-anxiety/Anti-panic agents; Anti-obsessive agents; Prescription stimulants (e.g., Provigil, Ritalin); Diet Pills/Anorectics; Systemic Steroids; Daily medication for chronic pain (e.g., opiates) or muscle spasms; Daily use of over the counter stimulants in pill form (e.g., ephedrine)
* Anti-coagulants (e.g., Warfarin)
* Any heart medications (e.g., dobutamine, isoproterenol)
* Daily medication for asthma
* Parkinson's disease medications (e.g., levodopa, methyldopa, apomorphine)
* Sympathomimetic (e.g., albuterol, pseudoephedrine)
* Other smoking cessation medications (Wellbutrin/Zyban, Chantix/varenicline)

Medical Exclusion Criteria:

* Women who are pregnant, planning a pregnancy within the next 3 months, or lactating.
* History or current diagnosis of any Axis 1 disorder as identified by the MINI (Mini International Neuropsychiatric Interview) or self-report. For major depression, only a current diagnosis will be exclusionary.
* History or current diagnosis of Attention-Deficit Hyperactivity Disorder (ADHD).
* Serious or unstable disease (e.g., cancer within the past 6 months [except squamous cell carcinoma], HIV, Parkinson's disease).
* History of epilepsy or a seizure disorder.
* History or current diagnosis (last 6-months) of abnormal rhythms and/or tachycardia (>100 beats/minute); history or current diagnosis of COPD, cardiovascular disease (stroke, angina, coronary heart disease); heart attack in the last 6 months; uncontrolled hypertension (SBP>150 or DBP>90).
* History or current kidney and/or liver failure (including transplant), disease, or impairment (e.g., cirrhosis); history or current diagnosis of hepatitis (excluding hepatitis A); liver function tests more than 20% outside of the normal range; Gamma-glutamyl Transpepsidase (GGT) values greater than 20% outside the normal range.
* Allergy to the study medication, tolcapone (Tasmar).
* History of severe, uncontrolled muscle movements (e.g., uncontrolled jerking, twitching) or a certain severe muscle problem (rhabdomyolysis).
* Low or borderline intellectual functioning - determined by receiving a score of less than 90 on the Shipley Institute of Living Scale (SILS) which correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated IQ Test (administered at the medical screening visit).
* Experience of dizziness or lightheadedness upon standing on a daily basis.
* Lifetime history of stroke.

fMRI Exclusion Criteria:

* Self-reported history of claustrophobia.
* Left-handedness.
* Color blindness.
* Any impairment preventing subjects from using response pad necessary for cognitive testing.
* Circumstances or conditions that may interfere with magnetic resonance imaging (MRI).
* Having a cochlear implant or wearing bilateral hearing aids.
* Self-reported history of head trauma (including being knocked unconscious for 3 minutes or greater and diagnosis of a concussion) or CNS tumor.
* Self-reported use of pacemakers, certain metallic implants, or presence of metal in the eye as contraindicated for MRI.
* History of gunshot wound.
* Weight greater than 300lbs. at medical screening or either testing day.
* Completion of cognitive testing in study #810493 or #811325 within the last 6 months.

Genetic Profile Exclusion Criteria:

* In order to balance the distribution of males and females, some participants who meet genotype and other eligibility criteria may not be enrolled in the study.

General Exclusion Criteria:

* Any medical condition or concomitant medication that could compromise subject safety or treatment, as determined by the Principal Investigator and/or Study Physician.
* Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, Ph.D., Principal Investigator — University of Pennsylvania; James Loughead, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in March 2010. Former study subjects with a known catechol-O-methyltransferase (COMT) genotype and who asked to be contacted for future studies were invited to participate, as well as potential subjects who called our center in response to advertising. All sessions were completed in our clinic at the University of Pennsylvania.
Pre-assignment Details: 2670 subjects completed initial screening over the phone; 669 (25%) were eligible. Of these, 418 (62%) scheduled an in-person screening visit; 218 (50%) attended this visit. 73 (17%) provided blood samples to determine final eligibility, based on genetic & liver function tests. 54 (74%) reached final eligibility; 46 (85%) started study medication.
Groups:
- Placebo First, Then Tolcapone: Subjects were asked to take study medication each day during two 11-day study medication periods. Between the two study medication periods was a washout period (no medication or visits) that lasted at least 10 days. During this washout period, subjects did not take any study medication and were asked to return to their normal smoking levels.
  Study medication assignment for each subject was randomized and counterbalanced, meaning approximately 50% of subjects took placebo during the first medication period, followed by tolcapone during the second medication period.
  During the placebo medication period, subjects followed a medication regimen and took capsules that were identical to those in the active tolcapone medication period (see protocol section for complete description).
- Tolcapone First, Then Placebo: Subjects were asked to take study medication each day during two 11-day study medication periods. Between the two study medication periods was a washout period (no medication or visits) that lasted at least 10 days. During this washout period, subjects did not take any study medication and were asked to return to their normal smoking levels.
  Study medication assignment for each subject was randomized and counterbalanced, meaning approximately 50% of subjects took tolcapone during the first medication period, followed by a placebo during the second medication period.
  During the active tolcapone medication period, subjects followed a tapered dosing schedule (see protocol section for complete description).
Period: Medication Period 1
Arm/Group | Placebo First, Then Tolcapone | Tolcapone First, Then Placebo
Started | 22 | 24
Completed | 18 | 17
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Ineligible: Positive Urine Drug Screen | 0 | 3
Not completed — Ineligible: fMRI contraindicated metal | 0 | 2
Not completed — Ineligible: Claustrophobia in fMRI | 2 | 0
Period: Washout Period
Arm/Group | Placebo First, Then Tolcapone | Tolcapone First, Then Placebo
Started | 18 | 17
Completed | 16 | 16
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: Medication Period 2
Arm/Group | Placebo First, Then Tolcapone | Tolcapone First, Then Placebo
Started | 16 | 16
Completed | 16 | 13
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: Measurements were taken during their first study visit, the medical screening visit.
Groups:
- Entire Study Population: Includes all subjects who were randomized to both study treatment groups (i.e., receive both placebo first and tolcapone first) and initiated study medication.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (12.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  African American | 15
  Caucasian | 29
  More than one race | 2
Region of Enrollment [Number; unit: participants]
  United States | 46
Nicotine Dependence [Mean (Standard Deviation); unit: Scores on a scale] — Determined by the Fagerstrom Test for Nicotine Dependence (FTND). The FTND is a 6-item, self-report measure of nicotine dependence derived from the Fagerstrom Tolerance Questionnaire. Scores range from 0-10; higher FTND scores indicate greater difficulty in quitting smoking. All subjects completed the FTND during the medical screening visit.
  Scores on a scale | 4.8 (1.5)
Cigarettes smoked per day [Mean (Standard Deviation); unit: Cigarettes smoked per day] — During the medical screening visit, subjects were asked to self-report the number of cigarettes they smoked on an average day.
  Cigarettes smoked per day | 17.1 (4.9)
Number of years smoked [Mean (Standard Deviation); unit: years] — During the medical screening visit, subjects were asked to self-report the number of years they have been a regular smoker (defined as smoking at least one cigarette per day).
  years | 21.8 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Measure of Brain Activity: Blood Oxygen Level Dependent (BOLD) fMRI Signal Change During the "N-back" Working Memory Task (Brain Region: Right Dorsolateral Prefrontal Cortex; Right DLPFC)
Description: Subjects completed two, 11-day study medication periods (one taking active tolcapone; one taking placebo). On Day 8 of each period, after at least 24 hours of smoking abstinence, subjects had an fMRI scan to measure changes in brain activity that occur during a memory test. The subjects completed a commonly used working memory test referred to as the "N-back". This test presented complex geometric figures on a projection screen for 0.5 seconds; each figure is separated by 2.5 seconds of black screen. There were 4 conditions requiring increasing memory demands: 0-back, 1-back, 2-back, & 3-back. Subjects had to respond to the target geometric figure that was separated by 0, 1, 2, or 3 figures before it is repeated. Between each condition, there was a brief rest period.
  To identify brain signal change, we calculated the difference in the amount of brain activity detected by the fMRI scan for each condition compared to the rest periods. This was a within-subject analysis.
Time Frame: At fMRI scan sessions - Days 8 and 29
Population: 29 subjects completed both fMRI scan sessions; however, data from 9 subjects were excluded from analysis, due to either poor fMRI data quality, low task accuracy (defined as task scores falling two standard deviations below the mean), or a failure to respond to more than 30% of the task's items. Below, we report on the 20 remaining subjects.
Measure: Mean (Standard Error); unit: BOLD signal
Groups:
- Placebo: An 11-day placebo-controlled medication period.
  Both medication periods involved taking identical capsules in the same tapered-dose regimen (Day 1: 100mg three times daily, Days 2-8: 200mg three times daily, Day 9: 200mg twice daily, Day 10: 200mg once daily, Day 11: 100mg once daily). The only difference was that, during the placebo period, the capsules did not contain tolcapone.
  All medication was encapsulated by the University of Pennsylvania's Investigational Drug Service (IDS).
- Tolcapone: 11-day medication period following a tapered dosing scheduled (Day 1: 100mg three times daily, Days 2-8: 200mg three times daily, Day 9: 200mg twice daily, Day 10: 200mg once daily, Day 11: 100mg once daily). The only difference was that, during this period, the capsules contained the active medication, tolcapone.
  All medication was encapsulated by the University of Pennsylvania's Investigational Drug Service (IDS)
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
BOLD signal | 0.27 (0.04) | 0.27 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that tolcapone would increase BOLD signal, meaning there would be an increase in brain activity, in the right dorsolateral prefrontal cortex, a part of the brain known to be involved in working memory. We analyzed for main effects of treatment (tolcapone vs. placebo), back level (0, 1, 2, and 3), treatment order, and relevant covariates (genotype, race, age, sex, FTND score, Shipley IQ score); Test type: Superiority or Other; p = 0.88, Regression, Linear — Because the five "a priori" brain regions of interest (ROIs) are highly correlated, the significance threshold was adjusted to p=0.014; BOLD signal change was examined using random effects maximum likelihood regression

2. Secondary Outcome: Cognitive Performance: Accuracy
Description: Subjects underwent two, 11-day study medication periods (one taking active tolcapone; one taking placebo). On Day 8 of each study medication period, after at least 24 hours of smoking abstinence, subjects completed an fMRI brain scan. During these fMRI scan sessions, participants completed computer tasks that were designed to test working memory and attention. These tasks were similar to computer games, in that participants would push a button in response to the pictures they see.
  Specifically, we tested whether subjects, while taking tolcapone, would display increased accuracy during the N-back working memory task compared to their performance while they took the placebo. We measured accuracy by counting the absolute number of true positives scored (the number each subject got correct during the task). This was a within-subject analysis.
Time Frame: At fMRI scan sessions - Days 8 and 29
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of true positives
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
Number of true positives | 49.9 (1.3) | 51.8 (0.87)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that tolcapone (vs. placebo) would increase subject's accuracy during the N-back working memory task; Test type: Superiority or Other; p = 0.017, Regression, Linear — The threshold for statistical significance was not adjusted. Significance remained at p=0.05; Accuracy was examined using random effects maximum likelihood regression

3. Secondary Outcome: Cognitive Performance: Reaction Time
Description: Subjects underwent two, 11-day study medication periods (one taking active tolcapone; one taking placebo). On Day 8 of each study medication period, after at least 24 hours of smoking abstinence, subjects completed an fMRI brain scan. During these fMRI scan sessions, participants completed computer tasks that were designed to test working memory and attention. These tasks were similar to computer games, in that participants would push a button in response to the pictures they see.
  Specifically, we tested whether subjects, while taking tolcapone, would display increased average reaction time (in milliseconds) during the N-back working memory task compared to their performance while they took the placebo. This was a within-subject analysis.
Time Frame: At fMRI scan sessions - Days 8 and 29
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
Milliseconds | 518 (16) | 520 (16)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that tolcapone (vs. placebo) would reduce subject's reaction time during the N-back working memory task; Test type: Superiority or Other; p = 0.88, Regression, Linear — The threshold for statistical significance was not adjusted. Significance remained at p=0.05; Examined using random effects maximum likelihood regression

4. Secondary Outcome: Subjective Symptoms: Smoking Behavior
Description: In order to determine if tolcapone (vs. placebo) would affect subject smoking behavior, we collected the daily number of cigarettes each subject smoked from Days 1 through 7 during each study medication period. This allowed us to calculate the average number of daily cigarettes smoked, across all subjects, during each study medication period (i.e., the average number of cigarettes/day smoked while all subjects took tolcapone and the average number of cigarettes/day smoked while all subjects took placebo). Then, we statistically assessed if there was a significant difference between these averages.
Time Frame: Days 1 through 7 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Average number of cigarettes smoked/day
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
Average number of cigarettes smoked/day | 14.2 (3.9) | 14.3 (4.0)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that smokers would smoke fewer cigarettes while taking tolcapone (vs. placebo); Test type: Superiority or Other; p = 0.85, Regression, Linear — The threshold for statistical significance was not adjusted. Significance remained at p=0.05; Examined using random effects maximum likelihood regression

5. Secondary Outcome: Subjective Symptoms: Cigarette Craving
Description: Subjective symptoms were assessed during each in-person session throughout each study medication period. During each visit, we asked subjects to complete the Questionnaire for Smoking Urges-Brief (QSU-B). Specifically, subjects completed the QSU-B at day 5, day 8 (fMRI scanning session 1), day 26 (day 5 of study medication period 2), and day 29 (day 8 of study medication period 2; fMRI scanning session 2).
  The range of possible scores on the QSU-B is 10-70, with higher values indicating an increased craving for cigarettes. This range of scores represent a "total" score; there are no subscales.
  While the QSU-B was collected at all in-person sessions, we only analyzed the scores collected from the fMRI scanning sessions of each period (day 8 and day 29). To analyze, we averaged the total scores across all 20 subjects from each fMRI scanning session and statistically analyzed for significant differences between these two averages. This was a within-subject analysis.
Time Frame: Day 8 (fMRI scanning session) of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
units on a scale | 40.5 (14.7) | 42.0 (12.6)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that smokers, while taking tolcapone (vs. placebo), would experience less cigarette craving during their 24-hour abstinence period; Test type: Superiority or Other; p = 0.40, Regression, Linear — The threshold for statistical significance was not adjusted. Significance remained at p=0.05; Examined using random effects maximum likelihood regression

6. Secondary Outcome: Subjective Symptoms: Withdrawal Symptoms
Description: Subjective symptoms were assessed during each in-person session throughout each study medication period. During each visit, we asked subjects to complete the Minnesota Nicotine Withdrawal Scale - Revised version (MNWS). The scale assesses eight DSM-IV items of nicotine withdrawal. The range of possible total scores on the MNWS is 0-60, with higher values indicating an increased nicotine withdrawal. This range of scores represent a "total" score; there are no subscales. The MNWS-N (right now/at the moment) was assessed during each fMRI scanning session visit (Day 8).
  To assess if tolcapone (vs. placebo) affect withdrawal symptoms, we statistically analyzed the average of the total MNWS scores across, all 20 subjects, for each study medication period. Specifically, we analyzed for significant differences between reported withdrawal symptoms while taking tolcapone vs. taking placebo.
Time Frame: Day 8 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo; Tolcapone: See "Protocol" or "Participant Flow" sections for full description of this study arm.
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
units on a scale | 10.9 (7.9) | 10.0 (7.7)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that smokers, while taking tolcapone (vs. placebo), would experience fewer withdrawal symptoms during their 24-hour abstinence period; Test type: Superiority or Other; p = 0.43, Regression, Linear — The threshold for statistical significance was not adjusted. Significance remained at p=0.05; Examined using random effects maximum likelihood regression

7. Primary Outcome: Measure of Brain Activity: Blood Oxygen Level Dependent (BOLD) fMRI Signal Change During the "N-back" Working Memory Task (Brain Region: Left Dorsolateral Prefrontal Cortex; Left DLPFC)
Description: as for outcome 1
Time Frame: At fMRI scan sessions - Days 8 and 29
Population: See previous sections.
Measure: Mean (Standard Error); unit: BOLD signal
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
BOLD signal | 0.32 (0.03) | 0.28 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that tolcapone would increase BOLD signal, meaning there would be an increase in brain activity, in the left dorsolateral prefrontal cortex, a part of the brain known to be involved in working memory. We analyzed for main effects of treatment (tolcapone vs. placebo), back level (0, 1, 2, and 3), treatment order, and relevant covariates (genotype, race, age, sex, FTND score, Shipley IQ score); Test type: Superiority or Other; p = 0.18, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; BOLD signal change was examined using random effects maximum likelihood regression

8. Primary Outcome: Measure of Brain Activity: Blood Oxygen Level Dependent (BOLD) fMRI Signal Change During the "N-back" Working Memory Task (Brain Region: Dorsal Cingulate/Medial Prefrontal Cortex; MF/CG)
Description: as for outcome 1
Time Frame: At fMRI scan sessions - Days 8 and 29
Population: See previous sections.
Measure: Mean (Standard Error); unit: BOLD signal
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
BOLD signal | 0.39 (0.03) | 0.37 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that tolcapone would increase BOLD signal, meaning there would be an increase in brain activity, in the dorsal cingulate/medial prefrontal cortex, a part of the brain known to be involved in working memory. We analyzed for main effects of treatment (tolcapone vs. placebo), back level (0, 1, 2, and 3), treatment order, and relevant covariates (genotype, race, age, sex, FTND score, Shipley IQ score); Test type: Superiority or Other; p = 0.67, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; BOLD signal change was examined using random effects maximum likelihood regression

9. Primary Outcome: Measure of Brain Activity: Blood Oxygen Level Dependent (BOLD) fMRI Signal Change During the "N-back" Working Memory Task (Brain Region: Posterior Cingulate Cortex; PCC)
Description: as for outcome 1
Time Frame: At fMRI scan sessions - Days 8 and 29
Population: See previous sections.
Measure: Mean (Standard Error); unit: BOLD signal
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
BOLD signal | -0.34 (0.05) | -0.33 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that tolcapone would increase suppression of BOLD signal, meaning an increase in suppression of brain activity, in the posterior cingulate cortex, a part of the brain known to be involved in working memory. We analyzed for main effects of treatment (tolcapone vs. placebo), back level (0, 1, 2, and 3), treatment order, and relevant covariates (genotype, race, age, sex, FTND score, Shipley IQ score); Test type: Superiority or Other; p = 0.98, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; BOLD signal change was examined using random effects maximum likelihood regression

10. Primary Outcome: Measure of Brain Activity: Blood Oxygen Level Dependent (BOLD) fMRI Signal Change During the "N-back" Working Memory Task (Brain Region: Ventromedial Prefrontal Cortex; vmPFC)
Description: as for outcome 1
Time Frame: At fMRI scan sessions - Days 8 and 29
Population: See previous sections.
Measure: Mean (Standard Error); unit: BOLD signal
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 20 | 20
BOLD signal | -0.29 (0.06) | -0.45 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Tolcapone; We hypothesized that tolcapone would increase suppression of BOLD signal, meaning an increase in suppression of brain activity, in the ventromedial prefrontal cortex, a part of the brain known to be involved in working memory. We analyzed for main effects of treatment (tolcapone vs. placebo), back level (0, 1, 2, and 3), treatment order, and relevant covariates (genotype, race, age, sex, FTND score, Shipley IQ score); Test type: Superiority or Other; p = 0.002, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; BOLD signal change was examined using random effects maximum likelihood regression

ADVERSE EVENTS:
Time Frame: A checklist of side effects was administered to subjects at the baseline session, day 5, day 8, day 26, and day 29, asking subjects if they experienced and to rate known side effects of tolcapone on a scale of "none," "mild," "moderate," "severe."
Description: Additionally, subjects were given instructions and contact information to call the study physician if they experienced severe side effects at any time. The study physician was consulted if moderate or severe side effects were reported, who would determine the severity and outcome of the AE.
Groups:
- Placebo: 11-day placebo-controlled medication period. Placebo capsules are identical to those in the active tolcapone treatment. When taking placebo, subjects follow an identical dosing schedule as the active treatment period.
  Placebo: Participants will be asked to take study medication each day for both 11-day study medication periods.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take tolcapone during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by tolcapone during the second medication period.
- Tolcapone: 11-day phase, tapered dosing scheduled (Day 1: 100mg three times daily, Days 2-8: 200mg three times daily, Day 9: 200mg twice daily, Day 10: 200mg once daily, Day 11: 100mg once daily); oral dosing; medication is encapsulated by the University of Pennsylvania's Investigational Drug Service (IDS)
  Tolcapone: Participants will be asked to take study medication each day for both 11-day study medication periods.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take tolcapone during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by tolcapone during the second medication period.
Arm/Group | Placebo | Tolcapone
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

LIMITATIONS AND CAVEATS:
Genetic studies, particularly imaging studies, have drawbacks such as small sample size and focus on single candidate genes; both can be said of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes